CLINICAL TRIAL: NCT05783570
Title: A Dose-escalation, Single-arm, Open-Label, Phase 1 Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of EU307, Autologous Glypican 3 Targeted Chimeric Antigen Receptor T Cell Therapy in Patients With GPC3 Positive Advanced Hepatocellular Carcinoma Who Have Failed Standard Therapy
Brief Title: To Evaluate the Safety, Tolerability and Preliminary Efficacy of EU307
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eutilex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-CTS307-I-01
Record Dates: First submitted 2023-02-27; First posted 2023-03-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: GPC3; HCC; Hepatocellular Carcinoma; CAR-T
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EU307 CAR-T Cell (Experimental)
  Interventions: Biological: EU307 CAR-T Cell

INTERVENTIONS:
Biological: EU307 CAR-T Cell — * Dose to be administered: a single dose
  * IV administration
  * Dosing rate: To be administrated at a rate of approximately 2 mL/min

SUMMARY:
To Evaluate the Safety, Tolerability and Preliminary Efficacy of EU307, Autologous Glypican 3 (GPC3) Targeted Chimeric Antigen Receptor T cell therapy in Patients with GPC3 Positive Advanced Hepatocellular Carcinoma who Have Failed Standard Therapy

DETAILED DESCRIPTION:
A Dose-escalation, Single-arm, Open-Label, Phase 1 Study

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, subjects must meet all of the following criteria:

  1. Male or female adults ≥19 years old at the time of written informed consent
  2. Patients with histologically or cytologically diagnosed unresectable HCC refractory to first- or second-line standard therapy* with no other standard therapy available

     * Including, but not limited to atezolizumab plus bevacizumab combination therapy and tyrosine kinase inhibitors (e.g., sorafenib, lenvatinib).
  3. Confirmed GPC3 positivity by IHC based on a liver tissue sample
  4. At least 1 measurable lesion based on mRECIST v1.1
  5. Child-Pugh score Class A or Class B(7)
  6. Life expectancy ≥3 months based on the judgment of the investigator
  7. ECOG PS 0 or 1
  8. Patients who have adequate bone marrow, liver, and kidney functions at the time of screening:

     WBC ≥ 2,000 /μL ANC ≥ 1,000 /μL Platelet ≥ 80,000 /μL Hemoglobin ≥ 9.0 g/dL Albumin ≥ 2.8 g/dL AST and ALT ≤ 5ⅹULN Total bilirubin ≤ 2 x ULN Serum creatinine ≤1.5 x ULN Creatinine clearance (CrCl) ≥ 30 mL/min PT(INR) ≤1.5 x ULN
  9. Negative serum pregnancy test in women of childbearing potential
  10. Women of childbearing potential or men who do not plan a pregnancy during the study period and who agree to use clinically adequate methods of contraception as follows:

      * Hormone contraceptives (subcutaneous implants, injections, oral contraceptives, etc.), intrauterine device (IUD) (or intra uterine system [IUS]), subject's or partner's surgical sterilization (vasectomy, tubal ligation, etc.), double barrier methods (combined use of barrier methods such as combined use of cervical cap or diaphragm plus male condom)
  11. Written informed consent to voluntary study participation

      Exclusion Criteria:
* Subjects who meet any of the following criteria cannot participate in the study:

Current disease and medical history

1. History or current evidence of hepatic encephalopathy
2. Patients with radiographic findings of brain metastases or spinal cord compression
3. Histologically confirmed HCC in ≥50% of the liver
4. Severe ascites requiring treatment such as paracentesis
5. History or current evidence of the following infections:

   * Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
   * Active hepatitis B (However, if HBsAg is positive, and if it is low or undetectable HBV DNA (HBV DNA level <2,000 IU/mL) based on the site-specific criteria at screening and a prophylactic antiviral agent can be administered for 6 months after the administration of the investigational product, enrollment is possible at the discretion of the investigator.)
   * Active hepatitis C (However, patients who have undergone antiviral therapy and whose HCV viral load is negative based on the site-specific criteria will be allowed to be enrolled.)
   * Uncontrolled severe chronic infection or active infection
6. Prior or planned organ transplantation during the study period
7. Diagnosis of any malignant tumor other than the study indication within 5 years prior to screening (Patients who were treated and assessed as complete response [CR] without recurrence within 3 years or patients diagnosed with nonmelanoma skin cancer, in-situ disease, thyroid cancer, or borderline tumor will be allowed to be enrolled.)
8. Clinically significant, severe cardiac disease based on the judgment of the investigator (e.g., uncontrolled hypertension, congestive heart failure [NYHA Grade ≥2], ventricular arrhythmia, active ischemic heart disease, history of myocardial infarction within 1 year prior to screening), renal impairment, or respiratory disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AEs (including DLT) | up to 6 month from LPI
  In this study, DLT is defined as an AE related to the IP (EU307),and severity will be assessed according to NCI-CTCAE v5.0
Production of replication competent lentiviruses (RCL) | up to 6 month from LPI
Development of anti-drug antibodies (ADA) | up to 6 month from LPI

SECONDARY OUTCOMES:
ORR | up to 6 month
  Proportion of subjects with confirmed CR or partial response (PR) as best overall response (BOR)
DoR | up to 6 month
  Time from confirmed tumor response (CR or PR) to confirmed progressive disease (PD)
DCR | up to 6 month
  Proportion of subjects with confirmed CR, PR, or stable disease (SD) (≥ 6 weeks) as BOR
TTR | up to 6 month
  Time from IP dosing to confirmed objective response (CR or PR)
TTP | up to 6 month
  Time from IP dosing to PD
PFS | up to 6 month
  Time from IP dosing to PD or all-cause death, whichever is earlier
OS | up to 6 month
  Time from IP dosing to all-cause death

OTHER OUTCOMES:
Quantitative CAR-T DNA assay | up to 6 month
Immunological assessment | up to 6 month
  -To explore relationship to tumor response, parameters to be analyzed include, but are not limited to: IFN-g, TNF-a, IL-2, IL-6, IL-18, IL-10, RANTES, MCP-1, TGF--Analysis of T cells and immune cells

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - National Cancer Center, Gyeonggi-do
  - Severance Hospital, Seoul
  - SoonChunHyang University Hospital Seoul, Seoul
  - The Catholic University of Korea Seoul ST.MARY'S Hospital., Seoul

IPD SHARING:
Plan to Share IPD: No